CLINICAL TRIAL: NCT03644472
Title: Postmenopausal Women and Their Endothelium: Is Dietary Nitrate Supplementation Protective
Brief Title: Postmenopausal Women and Their Endothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, David N. Proctor, PhD, Professor of Kinesiology, Physiology, and Medicine, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 00010017
Record Dates: First submitted 2018-08-20; First posted 2018-08-23 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Postmenopausal Women
Keywords: dietary nitrate supplementation; beetroot juice

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrate rich beetroot juice (Active Comparator): Subjects will consume 140 ml of beetroot juice (Beet-It Organic Shot) approximately 90 min before physiological testing.
  Interventions: Drug: nitrate rich beetroot juice
- Nitrate depleted beetroot juice (Placebo Comparator): Subjects will consume 140 ml of beetroot juice (Beet-It Organic Placebo) approximately 90 min before physiological testing.
  Interventions: Drug: nitrate depleted beetroot juice

INTERVENTIONS:
Drug: nitrate rich beetroot juice — This beverage contains 0.3 g of inorganic nitrate per 70 ml container, and is bottled and supplied by James White Drinks (UK).
  Other Names: Beet-It Organic Shot
  Arms: Nitrate rich beetroot juice
Drug: nitrate depleted beetroot juice — This beverage is identical in look and taste to the Beet-It organic shot, but has the nitrate removed. It is also bottled and supplied by James White Drinks (UK).
  Other Names: Beet-it Organic Shot Placebo
  Arms: Nitrate depleted beetroot juice

SUMMARY:
The purpose of this study is to test the effects of a one time dose and 7-days of inorganic nitrate (supplied in the form of beetroot juice) on blood vessel function and resting blood pressure in healthy, postmenopausal women. Participants will drink beetroot juice and a placebo juice on separate visits where blood pressure and blood vessel function will be measured.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in the United States. Due to the loss of estrogen, women experience a unique accelerated rise in cardiovascular disease risk factors following menopause. Postmenopausal women represent a population at heightened risk for cardiovascular disease development. Function of the endothelium has been shown to decline across the menopause transition, resulting in less production of nitric oxide. As such the investigators are investigating a potential therapeutic strategy in women have recently undergone menopause to boost nitric oxide availability.

ELIGIBILITY:
Inclusion Criteria:

* Early post-menopausal women who are within 1-6 years following their final menstrual cycle
* Late post-menopausal women who are beyond 6 years following their final menstrual cycle

Exclusion Criteria:

* Individuals with any overt cardiovascular, metabolic, hematologic, pulmonary, renal, musculoskeletal, and/or neurological disease(s).
* Users of any tobacco and/or nicotine products (smokers, chewing tobacco, nicotine-containing patches/gum, smokeless cigarettes)
* Individuals with a BMI > 35
* Individuals with resting blood pressure > or = 130/80 mm Hg
* Individuals with high blood lipids (total cholesterol > or = 240 mg/dl, LDL > or = 160 mg/dl, triglycerides > or = 200 mg/dl).
* Postmenopausal women with hyperglycemia (fasting glucose > or = 110 mg/dl and HbA1c >6.0%).
* Individuals taking any of the following medications:

  1. blood pressure lowering medication (e.g., beta blockers, ACE inhibitors, angiotensin antagonists, calcium channel blockers, diuretics)
  2. lipid- lowering medication (e.g., statins)
  3. nitrates (e.g. nitroglycerin) for angina
  4. phosphodiesterase inhibitors (e.g., Viagra)
  5. anti-Inflammatory drugs
* Individuals taking hormone therapy

Max Age: 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Postmenopausal women assigned as female at birth
Enrollment: 37 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Macro-vascular reactivity | These measurements will take place before and after a ischemia-reperfusion injury (20 minutes inflation, 20 minutes deflation) induced in the upper arm to assess change in macro-vascular reactivity
  Using near-infrared spectroscopy, a probe placed on the forearm muscle will be used to measure the tissue saturation index re-perfusion slope following 5 minutes of forearm cuff occlusion.
Micro-vascular reactivity | These measurements will take place before and after a ischemia-reperfusion injury (20 minutes inflation, 20 minutes deflation) induced in the upper arm to assess change in micro-vascular reactivity
  Using near-infrared spectroscopy, a probe placed on the forearm muscle will be used to measure area under the curve for tissue saturation index re-perfusion following 5 minutes of forearm cuff occlusion.

SECONDARY OUTCOMES:
Resting blood pressures | Change from baseline resting blood pressure and at 90 minutes after beet root juice ingestion
  Resting systolic blood pressures will be measured in the arm (cuff) and estimated in the aorta (radial artery tonometry).
Recovery of micro-vascular function and brachial artery flow mediated dilation | Change in these measures from immediately after ischemia-reperfusion injury to 30 minutes following
  Micro-vascular and brachial artery flow-mediated dilation, as described above, will be reassessed 30 minutes following ischemia-reperfusion injury to determine recovery of vessel function.
Brachial artery flow-mediated dilation | These measurements will take place before and after a ischemia-reperfusion injury (20 minutes inflation, 20 minutes deflation) induced in the upper arm to assess change in brachial artery flow-mediated dilation
  Using doppler ultrasound the brachial artery diameter will be measured before and after 5 minutes of forearm cuff occlusion
Brachial ankle pulse wave velocity and ankle-brachial index | These measurements will take place before (day 1) and 24 hours after (day 8) 7 days of supplementation.
  Using the VP-Colin 2000 brachial ankle pulse wave velocity and ankle brachial index will be measured before and after supplementation

CONTACTS AND LOCATIONS:
Overall Officials: David N Proctor, PhD, Principal Investigator — Penn State University
Locations (1):
- Penn State University, University Park, Pennsylvania, United States

REFERENCES:
- [Derived] Delgado Spicuzza JM, Gosalia J, Zhong L, Bondonno C, Petersen KS, De Souza MJ, Alipour E, Kim-Shapiro DB, Somani YB, Proctor DN. Seven-day dietary nitrate supplementation clinically significantly improves basal macrovascular function in postmenopausal women: a randomized, placebo-controlled, double-blind, crossover clinical trial. Front Nutr. 2024 Jun 10;11:1359671. doi: 10.3389/fnut.2024.1359671. eCollection 2024. PMID 38915856